CLINICAL TRIAL: NCT01904838
Title: The Healing Context in Complementary and Alternative Medicine (CAM): Instrument Development and Initial Validation - Calibration Study
Brief Title: The Healing Context in CAM: Instrument Development and Initial Validation - Calibration Study
Acronym: HEAL2
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Carol Greco, Assistant Professor of Psychiatry, University of Pittsburgh
Other Study IDs: AT006453 -2; R01AT006453 (NIH)
Record Dates: First submitted 2013-07-17; First posted 2013-07-22 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Persons Receiving Any Medical or Behavioral Treatment (Focus of Study is Questionnaires)

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Patients in Pittsburgh, Pennsylvania: persons receiving treatment at integrative and conventional medicine clinics in Pittsburgh, Pennsylvania
- Internet sample: internet sample of persons reporting that they receive, or have received in the past year, integrative medicine or conventional medical treatments.

SUMMARY:
The overall objective of this study is to develop and test an efficient set of self-report instruments to measure Complementary and Alternative Medicine(CAM)-relevant contextual factors important in healing. The initial phase of the study involves developing and refining an item bank. During the initial 'item bank development' phase, the investigators will run focus groups and cognitive interviews with individuals who participate in CAM and conventional medicine interventions. The next step of instrument development is called Calibration, and involves administering the revised item bank to an internet sample and to persons who receive services in a CAM clinic and a conventional primary care setting. The items will be calibrated using item response theory and classical test theory. This will result in a computerized adaptive testing version of the instrument, as well as a static short form of the instrument. This current protocol in ClinicalTrials.gov pertains only to the Calibration Phase of the study. The final phase of the project will involve conducting initial validation studies of the set of instruments. The set of instruments will be called the Healing Encounters and Attitudes Lists (HEAL). The investigators will evaluate the convergent, discriminant, and predictive validity of the HEAL instruments in a sample of 200 persons with chronic low back pain who are receiving physical therapy, chiropractic care, or mindfulness-based stress reduction. For convergent validity, the HEAL is expected to display moderate to large correlations with measures of similar constructs. The HEAL is expected to correlate modestly with self-report measures of general psychosocial functioning, in support of discriminant validity. Finally, HEAL scores should account for a significant proportion of the variance in treatment outcome, supporting predictive validity.

DETAILED DESCRIPTION:
This project will develop and test a set of patient self-report measurement tools to assess the perceived contextual factors, such as patient attitudes and expectations, patient provider relationship factors, and environmental factors that contribute to healing. Our project is synergistic with the National Institutes of Health (NIH) Roadmap initiative, Patient Reported Outcomes Measurement Information System (PROMIS), and will use the rigorous instrument development and validation methodology of PROMIS. The overall objective of this study is to develop efficient self-report instruments to measure CAM-relevant contextual factors important in healing, hereafter referred to as the Healing Encounters and Attitudes Lists (HEAL), and conduct initial validation in persons seeking CAM and conventional treatment for pain. Specific Aim 1: Develop an item bank. We will employ several iterative steps used successfully in PROMIS to identify items that assess contextual factors of healing relevant to CAM. Initial steps in developing an item bank include: a) compilation and evaluation of existing instruments and relevant questions, b) consultation with experts, and c) focus groups with individuals who participate in CAM and conventional medicine interventions, and d) item editing. During the initial year of this study, we expect to identify conceptual areas of potential importance to CAM interventions and patients, and identify and edit items to create an item bank assessing these conceptual areas. Specific Aim 2: Calibrate items. We will use item response theory (IRT) and classical test theory (CTT) to calibrate the items from Aim 1 on three samples: 1) an internet-based sample (n= 1400), 2) 125 outpatients participating in CAM interventions at our Center for Integrative Medicine (CIM), and 3) 125 outpatients at a General Internal Medicine clinic. During year 2-3 we administer the items in the item bank to the 1650 persons, conduct IRT and CTT analyses and refine the item bank to only those items that best assess the constructs. Specific aim 2 will result in a Computerized Adaptive Testing (CAT) version of the HEAL, which maximizes information while minimizing patient time burden. A static short form of the HEAL will be derived from the HEAL CAT in Aim 2. Specific Aim 3: Conduct initial validation studies. We will evaluate convergent, discriminant, and predictive validity of the Healing Encounters and Attitudes List (HEAL) in a sample of chronic low back pain (CLBP) patients receiving CAM and conventional medicine treatments. The validity studies will use two samples of adults with CLBP: 100 persons receiving CAM treatments: chiropractic manipulation (CM) or mindfulness-based stress reduction (MBSR) at the CIM, and 100 persons receiving conventional care (physical therapy) at Centers for Rehab Services referred by the General Internal Medicine Clinic (GIMC) of the University of Pittsburgh Medical Center (UPMC). We will administer the CAT version of the HEAL questionnaire developed in aims 1 and 2 as well as conventional measures of treatment expectancy, confidence in treatment provider, psychosocial functioning, and treatment outcome measures for CLBP of pain and disability. • Hypothesis 3a: Scores on the HEAL measure will display moderate to large correlations (r's > .50) with similar self-report measures, supporting convergent validity. • Hypothesis 3b: Scores on the HEAL measure will correlate modestly (r's = .20-.35) with self-report measures of general psychosocial functioning, supporting discriminant validity. • Hypothesis 3c: HEAL scores will account for a significant proportion of variance in treatment outcome in both samples. In addition, we predict that HEAL scores will demonstrate incremental validity, i.e., they will account for significant incremental variance in outcome beyond that accounted for by existing measures of treatment expectancy and related constructs.

ELIGIBILITY:
Inclusion Criteria:

* 1. age 18 or over
* 2. Males and Females
* 3. able to read, speak and understand English
* 4. able to complete informed consent procedures
* 5. able to complete questionnaires on a computer
* 6. (local sample arm:) began treatment within the past 4 weeks at the UPMC Center for Integrative Medicine or conventional medical clinics at UPMC.
* 7. (internet sample arm) self report of current or past year integrative medicine or conventional medical treatment.

Exclusion Criteria:

* 1. self reported History of schizophrenia or current psychotic symptoms
* 2. self reported uncontrolled current bipolar disorder
* 3. self report of substance dependence within the past 6 months
* 4. self reported history of organic neuropsychiatric syndromes (e.g., Alzheimer's, Parkinson's, dementia)
* 5. Lack of willingness or ability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Local clincal sample is persons receiving treatment at UPMC clinics or UPMC Center for Integrative Medicine.
  Internet sample is persons reporting current or past year conventional or integrative medicine treatment.
Sampling Method: Non-Probability Sample
Enrollment: 1650 (Actual)
Dates: Start 2012-09; Primary Completion 2013-09 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Patient-reported perspectives on relationship with provider, treatment expectancy, attitudes towards healthcare | Baseline (generally same day as enrollment, but may occur at a single study visit within 4 weeks of enrollment)
  Participants' opinions regarding factors that contribute to healing, such as important patient characteristics, provider characteristics, and environmental factors

CONTACTS AND LOCATIONS:
Overall Officials: Carol M Greco, Ph.D., Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Result] Greco CM, Yu L, Johnston KL, Dodds NE, Morone NE, Glick RM, Schneider MJ, Klem ML, McFarland CE, Lawrence S, Colditz J, Maihoefer CC, Jonas WB, Ryan ND, Pilkonis PA. Measuring nonspecific factors in treatment: item banks that assess the healthcare experience and attitudes from the patient's perspective. Qual Life Res. 2016 Jul;25(7):1625-34. doi: 10.1007/s11136-015-1178-1. Epub 2015 Nov 12. PMID 26563249